CLINICAL TRIAL: NCT03573063
Title: Starvation Effect on Androgen Metabolism in Healthy Young Women.
Brief Title: Studying the Starvation Effect on Androgen Metabolism in 20 Healthy Young Women and Comparison to Women With PCOS.
Acronym: SEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-00982
Record Dates: First submitted 2018-03-02; First posted 2018-06-29 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: PCOS Disease
Keywords: starvation; androgens; healthy women; PCOS
MeSH Terms: conditions — Starvation

STUDY DESIGN:
Intervention Model Description: Clinical study with biological sampling in healthy young women being nutrionally restricted (using encoded data)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Androgen metabolism after starvation (Other): Metabolism changes after 48 hours starvation in healthy women
  Interventions: Other: Androgen metabolism after starvation

INTERVENTIONS:
Other: Androgen metabolism after starvation — The 20 women will all undergo the same process of starvation for 48 hours. During this time three blood samples and three 24-hours urine samples will be collected. At baseline, the investigators will draw blood, perform a pregnancy test and collect the 24 hours urine as well as a spot urine.
  Then the 48 hours starvation starts and two blood and two 24 hours urine samples and spot urines will be collected after 24 and 48 hours in the morning. After the third visit the study is completed for the participant.

SUMMARY:
In this study, the investigators wanted to investigate the energy homeostasis and the steroid metabolism of 20 healthy, young and normal weight women aged between 16-35 years before and after a 48 hours fasting period.

The following substrates and hormone concentrations representing the carbohydrate, fat and protein metabolism will be measured from plasma or urine before and after fasting: glucose, insulin, lactate, alpha-synucleine, free fatty acids, beta-hydroxybutyrate (ketone bodies), carnitine (surrogate for acetyl-CoA) and alanine (amino acids). In addition, the investigators will measure 67 steroid metabolites by GC/MS and Biokrates AbsolutIDQ Steroid Assay in all collected urines and blood samples.

In the analysis of the data, the investigators will focus on correlations between biochemical parameters of the energy metabolism and parameters of the steroid metabolism, specifically the androgens. In addition, the steroid profiles obtained from healthy young women before and after fasting will be compared to steroid profiles of PCOS women in search for specific differences.

DETAILED DESCRIPTION:
The first aim of this study is to investigate the energy homeostasis and the steroid metabolism of healthy, young and normal weight women aged 16-35 years, before and after a 48 hours fasting period. Furthermore, second aim of this study is the comparison of their steroid profiles with PCOS women in search for specific differences.

In fact it might be therefore hypothesized that the energy metabolism in PCOS women functions like under (glucose) starvation conditions. In a pilot experiment performed in a healthy young women of normal weight, the investigators observed that short term starvation over 48 hours changed her steroid profile from normal to PCOS-like with elevated testosterone with elevated testosterone, DHT and androsterone/etiocholanolone ratio. It has been suggested that during normal fasting and feeding metabolic signals such as AMP/NAD+ and acetyl-CoA translate the energy state into specific metabolic programs. The investigators suggest that androgen biosynthesis might be one of these programs. Therefore, becoming hyperandrogenic during short term starvation might be normal, and the regulation between energy balance and androgen biosynthesis might be visible in healthy subjects, thereby hinting pathways leading to PCOS and better treatment options.

In this study the investigators will recruit 20 healthy, normal weight women aged 16-35 years with regular cycle and without drug treatment, including hormonal contraception. Characteristics of the participant and written informed consent with the study will be collected. The study will start 14-21 days after the last menstrual period of the participant. Twenty-four hours prior the first study visit the participant will collect a 24 hours urine sample and a spot urine.

On day one of the study, the participant will come early morning for the first visit to the Inselspital Bern. The participant will be informed again and the exact study protocol will be explained to make sure the participant is willing to fulfil the study requirements. The investigators will draw blood, perform a pregnancy test and collect the 24 hours urine as well as a spot urine. At this point the starvation period will start (=intake to a maximum of 500-800 kcal/d for 24 hours, depends on the weight of the participant). A dietary plan is provided by Mrs. T. Zürcher, Pediatric Dietician, Childrens' Hosp. Inselspital Berne.

This regimen is selected on the basis that the human body switches into a state of "hunger" and starts to burn fat instead of glucose after about 12 hours. During a 48 hours fasting period the metabolism changes dramatically. During this state hormonal and chemical changes will be investigated in blood and urine samples. During the starvation the participants have to stick strictly to the dietary restriction regimen, which they will monitor themselves. If the participants fails to do so, they will be excluded from continuation of the study and cannot participate a second time. Fasting state and thus compliance are visible in the measured lab data (e.g. ketone bodies).

Two blood samples and two 24 hours urine samples and spot urines will be collected after 24 and 48 hours in the morning. After the third visit the study is completed for the participant. The blood samples and urine samples will be stored at -20°C until the day of measurement. If agreed by the participant, data and samples will be used for future studies in the same research field.

The collected samples of the participant (three blood and three 24-hours urine samples) will be analysed for metabolic markers (glucose, potassium, insulin, lactate, free fatty acids, ketone-bodies (beta-hydroxy-butyrate), carnitin, alanin) and for a multitude of steroids (progesterons, androgens, estrogens, corticosterones, mineralocorticoids, glucocorticoids). The measurements will be conducted according to GLP-standards. All laboratory parameters will be analysed in the University Hospital of Berne (Inselspital) in the laboratories of the Institute of Clinical Chemistry and Steroid Laboratory of Nephrology.

The obtained data will be entered in an existing RedCap database established for PCOS research of the PI. Laboratory data will be statistically analysed and compared to previous data obtained from a currently closing PCOS study being analysed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-35
* Normal weight
* Healthy
* Postpubertal
* No drug treatments (including oral/hormonal anticonception)
* Informed consent

Exclusion Criteria:

* Hormone treatment (i.e.: hormonal contraception, cortisol)
* Hormone disorders
* Infertile
* Anorexic
* Obese
* Pregnant
* Chronic diseases

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome is changes in androgen metabolism. The evaluation will compare the steroid concentrations at the three time points with uni- and multivariate data analysis to detect fasting-related differences. | One year
  With GC/MS (urine) and LCMSMS (blood) 40 steroids in urine (ug/24h) and 18 steroids in serum (pg/ml or nmol/L) (Biokrates) will be measured; these includes Progesterones, Androgens, Estrogens, Corticosterones, Mineralocorticoids, Glucocorticoids. Other markers consist of glucose (mmol/L), potassium (mmol/L), insulin (mU/L), lactate (mmol/L), free fatty acids (umol/L), ketone-bodies (beta-hydroxy-butyrate), carnitin, alanin - all umol/L). All parameters will be analysed in the laboratories of the Institute of Clinical Chemistry and Steroid Laboratory of Nephrology of Inselspital. For more details please see list in Appendices of the Clinical Study Protocol (Page 38-41). All data are assessed as absolute values and follow-up is studied for changes in values rather than for normative values, which mostly do not exist for fasting intervention.

SECONDARY OUTCOMES:
Steroid profiles | One year
  Working hypothesis: Starvation may change steroid profiles in similar direction as PCOS? - To test this hypothesis the collected biological samples of the participant will be analysed for steroid metabolic markers (see primary outcome measures) to same markers collected from a cohort of PCOS women available from a previous study for comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Christa Flück, Principal Investigator — Pädiatrische Endokrinologie, Inselspital
Locations (1):
- Benjamin P. Magyar, Aarau, Switzerland